CLINICAL TRIAL: NCT04907799
Title: Daily Caloric Restriction in Overweight and Obese Adults With ADPKD
Brief Title: Daily Caloric Restriction in ADPKD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-2999; R01DK129259 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-06-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Dominant Polycystic Kidney; Overweight and Obesity
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Caloric Restriction (Experimental): The daily caloric restriction group will participate in a 2-year, group-based, behavioral weight loss intervention based on a 30% reduction in caloric intake and increased physical activity.
  Interventions: Behavioral: Daily caloric restriction
- Standard Advice Control (Other): The standard advice control group will receive an initial consultation with a registered dietician regarding current clinical recommendations for ADPKD without subsequent counseling sessions.
  Interventions: Other: Standard advice control

INTERVENTIONS:
Behavioral: Daily caloric restriction — Weight loss based on daily caloric restriction and increased physical activity
  Arms: Daily Caloric Restriction
Other: Standard advice control — Initial nutrition consultation without subsequent counseling
  Arms: Standard Advice Control

SUMMARY:
This clinical trial will determine whether a daily-caloric restriction-based weight loss intervention can slow kidney growth in adults with autosomal dominant polycystic kidney disease who are overweight or obese. The study will also evaluate changes in abdominal fat by magnetic resonance imaging. Blood and fat samples will provide insight into biological changes that may contribute to any observed benefits of the intervention.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is characterized by development and continued growth of numerous fluid-filled renal cysts that ultimately result in renal failure. Similar to the general population, the prevalence of overweight and obesity have been rising in ADPKD patients, effecting about two-thirds of individuals. Adipocytes do not simply act as a fat reservoir, but are active endocrine organs that promote release of pro-inflammatory cytokines, and thus, may be a promising clinical target for ADPKD management. Mounting evidence also suggests that a metabolic defect exists in ADPKD, which likely contributes to cystic epithelial proliferation and subsequent cyst growth. Additionally, the investigators recently reported that overweight and obesity are strong independent predictors of more rapid kidney growth. Collectively, these data suggest that interventions to reduce abdominal adiposity may slow ADPKD progression.

Initial results from the investigators' R03-funded pilot and feasibility study support that a 12-month daily caloric restriction (DCR)-based behavioral weight loss intervention in adults with ADPKD and overweight or obesity: 1) is feasible and acceptable; 2) slowed kidney growth (annual %∆ in height-adjusted TKV [htTKV]), which was highly correlated with weight loss; 3) reduced abdominal adiposity; and 4) altered pathways implicated in ADPKD progression and metabolism. These initial results suggest that a DCR-based behavioral weight loss intervention offers a promising strategy to slow ADPKD progression. However, the pilot and feasibility study was limited by a small sample size, relatively short duration, and lack of a control group. Thus, to translate these promising results of the pilot study towards clinical practice, the investigators are conducting a randomized, controlled clinical trial in a larger number of adults with ADPKD and overweight or obesity to directly compare the efficacy of a DCR-based behavioral weight loss intervention compared to control for slowing kidney growth (primary outcome) over a longer duration. Changes in abdominal adiposity will serve as a secondary outcome and effects of weight loss on circulating and adipose markers of biological pathways will provide mechanistic insight.

In a subset of participants recruited for this clinical trial, we will measure change in kidney oxidative metabolism, insulin sensitivity, plasma metabolomics, and gut microbiota. These additional measures will aim to compare kidney oxidative metabolism, insulin sensitivity, plasma metabolome and gut microbiota at baseline and 2 years. In addition, the investigators aim to define the relations among changes in kidney oxidative metabolism, insulin sensitivity, plasma metabolome, gut microbiota, total kidney volume, and body weight over 2 years. Currently, it is unknown if weight loss via DCR modifies renal energy expenditure, substrate utilization, plasma metabolomics, or the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* ADPKD diagnosis based on the modified Pei-Ravine criteria
* Body-mass index of 25-45 kg/m^2
* Estimated glomerular filtration rate ≥ 30 mL/min/1.73m^2
* Total kidney volume (htTKV) > 600 mL, calculated/estimated from a previous kidney ultrasound or magnetic resonance imaging
* Access to the internet with video chat capabilities
* No plans for extended travel (>2 weeks) without internet access during the 12-month intensive period
* Not currently participating in or planning to participate in any formal weight loss or physical activity program, or another interventional study
* Ability to provide informed consent

Exclusion Criteria:

* Diabetes mellitus
* Current smokers or history of smoking in the past 12 months
* Alcohol dependence or abuse
* History of hospitalization or major surgery within the last 3 months
* Untreated dyslipidemia
* Uncontrolled hypertension
* Pregnancy, lactation, or unwillingness to use adequate birth control
* Cardiovascular disease, peripheral vascular disease, or symptoms suggestive of cardiovascular disease: chest pain, shortness of breath at rest or with mild exertion, syncope
* Abnormal resting electrocardiogram (ECG): serious arrhythmias, including multifocal premature ventricular contractions (PVC's), frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, QTc interval > 480 msec or other significant conduction defects
* Significant pulmonary disease including: chronic obstructive pulmonary disease, interstitial lung disease, cystic fibrosis, or uncontrolled asthma
* Regular use of prescription or over-the-counter medications that may affect weight, appetite, food intake, or energy metabolism unless weight stable
* History of clinically diagnosed eating disorder including: anorexia nervosa, bulimia, binge eating disorder
* Weight loss of >5% in the past 3 months for any reason except post-partum weight loss; weight gain >5% requires assessment by PI
* Major psychiatric disorder (e.g., psychosis, schizophrenia, mania, bipolar disorder) or current severe depression, based on DSM-IV-TR criteria for Major Depressive Episode, which in the opinion of the Study MD would interfere with ability to adhere to dietary interventions)
* Inability to cooperate with or clinical contraindication for magnetic resonance imaging, including: severe claustrophobia, implants, devices, or non-removable body piercings
* Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in height-Adjusted Total kidney volume | Baseline, 24-months
  To assess kidney growth, we will measure height-adjusted total kidney volume by magnetic resonance imaging at baseline and 24 months to determine annual percent change.

SECONDARY OUTCOMES:
Change in abdominal adiposity | Baseline, 24-months
  Abdominal adiposity (subcutaneous, visceral, and total) will be assessed by magnetic resonance imaging.
Change in the ratio of insulin-like growth factor-1 (IGF-1)/ to GF binding protein-1 | Baseline, 12-months, 24-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in adiponectin (circulating) | Baseline, 12-months, 24-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in leptin (circulating) | Baseline, 12-months, 24-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in interleukin-6 (circulating) | Baseline, 12-months, 24-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in tumor necrosis factor-alpha (circulating) | Baseline, 12-months, 24-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in C-reactive protein (circulating) | Baseline, 12-months, 24-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in peripheral blood mononuclear cell protein expression of pAMPK/AMPK | Baseline, 12-months, 24-months
  PBMCs will be isolated from whole blood to assess protein expression
Change in peripheral blood mononuclear cell protein expression of pS6K/S6K | Baseline, 12-months, 24-months
  PBMCs will be isolated from whole blood to assess protein expression
Change in adiponectin (adipose tissue) | Baseline, 24-months
  A subcutaneous adipose tissue biopsy will be performed for assessment of this mechanistic biomarker.
Change in leptin (adipose tissue) | Baseline, 24-months
  A subcutaneous adipose tissue biopsy will be performed for assessment of this mechanistic biomarker.
Change in interleukin-6 (adipose tissue) | Baseline, 24-months
  A subcutaneous adipose tissue biopsy will be performed for assessment of this mechanistic biomarker.
Change in tumor necrosis factor-alpha (adipose tissue) | Baseline, 24-months
  A subcutaneous adipose tissue biopsy will be performed for assessment of this mechanistic biomarker.
Change in renal oxygen consumption | Baseline, 24-months
  Renal oxygen consumption will be assessed by a PET/CT scan using 11-C acetate in a sub-set of participants
Change in gut microbiota | Baseline, 24-months
  16S rRNA gene sequencing will be used for taxonomic characterization of the gut microbiota in a subset of participants.
Change in plasma metabolome | Baseline, 24-months
  Untargeted plasma metabolomics will be performed using high-performance liquid chromatography-tandem mass spectrometry in a subset of participants.

OTHER OUTCOMES:
Safety (adverse events) | 24-months
  Number of participants with treatment-related adverse events in each group as evaluated by the DSMB
Change in dietary Energy Intake | Baseline, 1-, 6-, 12-, and 24-months
  Multiple pass 24-hr dietary recalls will be analyzed to evaluate self-reported energy intake
Adherence | 24 months
  Self-reported dietary adherence using a 1-10 likert scale (10 is highest adherence)
Tolerability (dropout due to adverse events) | 24 months
  Subject dropout due to treatment-emergent adverse events
Change in free-living physical activity | Baseline, 6-, 12- and 24-months
  Estimated energy expenditure (METs) over a 7-day period will be quantified using the activPAL3 micro.
Change in percent body fat | Baseline, 24-months
  Percent body fat will be assessed via DEXA scan in a sub-set of participants.
Change in plasma choline | Baseline, 24-months
  Plasma choline will be analyzed by high-performance liquid chromatography-tandem mass spectrometry in a sub-set of participants.
Change in plasma trimethylamine | Baseline, 24-months
  Plasma trimethylamine will be analyzed by high-performance liquid chromatography-tandem mass spectrometry in a sub-set of participants.
Change in plasma trimethylamine-N-oxide | Baseline, 24-months
  Plasma trimethylamine-N-oxide will be analyzed by high-performance liquid chromatography-tandem mass spectrometry in a sub-set of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Nowak, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in ADPKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Cortinovis M, Perico N, Remuzzi G. The Need for Novel Therapeutic Directions in Autosomal Dominant Polycystic Kidney Disease Patient Care. Clin J Am Soc Nephrol. 2025 Dec 5. doi: 10.2215/CJN.0000000975. Online ahead of print. PMID 41348481
- [Derived] Nowak KL, Copeland TP, Ku E, Sarnak MJ, Gitomer B, Abebe KZ, Chapman A, Perrone R, Rahbari-Oskoui FF, Steinman T, Yu ASL, Chonchol M. Overweight Status, Obesity, and Progression to ESKD in Patients with Autosomal Dominant Polycystic Kidney Disease. Clin J Am Soc Nephrol. 2025 Apr 1;20(4):520-528. doi: 10.2215/CJN.0000000640. Epub 2025 Feb 19. PMID 39970002
- [Derived] Chebib FT, Nowak KL, Chonchol MB, Bing K, Ghanem A, Rahbari-Oskoui FF, Dahl NK, Mrug M. Polycystic Kidney Disease Diet: What is Known and What is Safe. Clin J Am Soc Nephrol. 2024 May 1;19(5):664-682. doi: 10.2215/CJN.0000000000000326. Epub 2023 Sep 20. PMID 37729939